CLINICAL TRIAL: NCT03276377
Title: Use of Vitamin K Antagonist and Neurocognitive Disorders in Older Adults : a Retrospective Study With Exposed and Non-exposed Groups
Brief Title: VItamin K Inhibition and NeurocoGnition (VIKING)
Acronym: VIKING
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017/19
Record Dates: First submitted 2017-09-04; First posted 2017-09-08 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Neurocognitive Disorders
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed to VKA: VKA intake Patients who have been taking VKA for at least 3 months
- Non-exposed to VKA: DOAC intake Patients who have been taking DOAC for at least 3 months

SUMMARY:
The primary objective of this study is to determine whether patients usually taking Vitamin K Antagonists (VKAs) exhibit a poorer global cognitive performance than control patients (matched on age, gender and indication for anticoagulation) taking direct oral anticoagulants (DOACs).

The secondary objectives are:

* to determine whether patients usually taking VKAs are more likely to have moderate to severe cognitive disorders than matched controls taking DOACs.
* to determine whether VKAs intake is associated with poorer executive functions.
* to determine on CT scans whether the VKAs intake is associated with a greater volume of vascular calcifications in the brain compared to the use of DOACs.

DETAILED DESCRIPTION:
VKAs are the most common drugs in the treatment and prophylaxis of thromboembolic events in older adults. Their action is mediated by decrease in the bioavailability of the active form of vitamin K. However, vitamin K participates in brain health and function by regulating the synthesis of sphingolipids, a constituent of the myelin sheath and the neurons membrane, and through the biological activation of vitamin K-dependent proteins (VKDPs) involved in neuron survival. Epidemiological studies have reported a positive association between higher serum vitamin K concentration and better verbal episodic memory performance in older adults, and an inverse association between dietary vitamin K intakes and cognitive complaint/cognitive disorders/behavioral disorders. VKAs, which deplete the active form of vitamin K, may thus be responsible for neurological disorders. CNS abnormalities were observed in newborns exposed in utero to VKA. Similarly, in two cross-sectional studies, the use of VKAs was directly associated with cognitive disorders in older adults, and with a lower volume of gray matter in the hippocampus.

However, the main limitation of these previous studies was that the different associations reported may actually be explained by the thromboembolic pathology justifying the use of VKA such as atrial fibrillation with potential adverse consequences on the brain.

Thus, the use of DOACs could serve as an ideal comparator, as their indications are similar to those of VKAs but which mechanism does not interfere with vitamin K.

The investigators hypothesize that 1) geriatric patients usually taking VKAs may have lower cognitive performance than those usually taking DOACs; 2) there is an association between VKA intake and cognitive performance in geriatric patients, including after adjustment on the indication for anticoagulation; and 3) that geriatric patients usually taking VKAs exhibit brain changes compared to those usually taking DOACs, including greater calcification burden.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years and over
* To be seen in consultation or day hospital in the department of geriatrics from 01/01/2015 to 31/12/2016
* Exposed :

  * Patients who have been taking VKA for at least 3 months for atrial fibrillation or pulmonary embolism, with INR between 2 and 3
* Non-exposed:

  * Patients who have been taking DOAC for at least 3 months for atrial fibrillation or pulmonary embolism
  * Matched on age (± 5 years), gender and indication for anticoagulation

Exclusion Criteria:

* Severe kidney failure (creatinine clearance < 30 mL/min)
* Language other than French

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients are recruited in the memory clinic and geriatric day hospital of the University Hospital of Angers, France
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of the global cognitive performance between geriatric patients exposed and non-exposed to VKA | Baseline
  Global cognitive performance is assessed by the Mini-Mental State Examination (MMSE) score

SECONDARY OUTCOMES:
Comparison of moderate-to-severe dementia diagnosis between geriatric patients exposed and non-exposed to VKA | Baseline
  Moderate-to-severe dementia defined as a MMSE score < 20 / 30
Comparison of the executive functions between geriatric patients exposed and non-exposed to VKA | Baseline
  Executive functioning is assessed by the Frontal Assessment Battery (FAB) score
Evaluation of the volume of vascular calcifications in the brain according to the use of VKAs | Baseline
  Semi-automated measure of the volume of vascular calcifications in the brain based on CT scan

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University Hospital, Angers, France